CLINICAL TRIAL: NCT00623428
Title: A Randomized, Open-label Study of the Effects of 24 vs 48 Weeks of Combination Therapy With PEGASYS (Peginterferon Alfa-2a 40KD) Plus COPEGUS (Ribavirin) on Sustained Virological Response in Patients With Chronic Hepatitis C, Genotype 2 or 3 Who do Not Achieve a Rapid Viral Response
Brief Title: A Study of Combination Therapy With PEGASYS (Pegylated Interferon Alfa-2a (40KD)) and Copegus (Ribavirin) in Patients With Chronic Hepatitis C Genotype 2 or 3 Who Do Not Achieve a Rapid Viral Response
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MV21371; 2007-004993-15
Record Dates: First submitted 2008-02-18; First posted 2008-02-26 (Estimated); Results first posted 2013-06-24 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

ARMS (2):
- PEG-IFN alfa-2a + Ribavirin for 24 weeks (Experimental): After 24 weeks of treatment with pegylated interferon alfa-2a (PEG-IFN alfa-2a) 180 μg/week plus ribavirin 800-1200 mg/day participants who achieved at least a 2-log10 drop of hepatitis C virus (HCV) ribonucleic acid (RNA) at Week 12 (as compared to HCV RNA levels prior to treatment initiation) or had HCV RNA <15 IU/mL, and who were still taking study medication at treatment Week 24 were randomized into the study, at which time treatment was stopped. Participants were followed for an additional 48 weeks during the treatment-free follow-up period.
  Interventions: Drug: peginterferon alfa-2a; Drug: Ribavirin
- PEG-IFN alfa-2a + Ribavirin for 48 weeks (Active Comparator): After 24 weeks of treatment with PEG-IFN alfa-2a 180 μg/week plus ribavirin 800-1200 mg/day participants who achieved at least a 2-log10 drop of HCV RNA at Week 12 (as compared to HCV RNA levels prior to treatment initiation) or had HCV RNA <15 IU/mL, and who were still taking study medication at treatment Week 24 were randomized into the study, and continued treatment for another 24 weeks (for a total of 48 weeks of treatment). Participants were followed for an additional 24 weeks during the treatment-free follow-up period.
  Interventions: Drug: peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: peginterferon alfa-2a
  Other Names: Pegasys®; PEG-IFN alfa-2a
Drug: Ribavirin
  Other Names: Copegus®

SUMMARY:
This study will evaluate the efficacy and safety of peginterferon alfa-2a 40KD + ribavirin combination therapy given for 24 weeks versus 48 weeks in patients with chronic hepatitis C, genotype 2/3.

DETAILED DESCRIPTION:
During a pre-study run-in phase patients with chronic hepatitis C genotype 2/3, who had started therapy with PEG-IFN alfa-2a plus ribavirin according to local standard of care and did not achieve a rapid viral response (RVR) (defined as Hepatitis C virus (HCV) RNA <15 IU/mL at Week 4 of treatment measured with the Roche COBAS AmpliPrep / COBAS TaqMan® HCV Test) were eligible for the study and entered the screening phase between treatment Week 4 and 8 as soon as the result of the Week 4 HCV RNA test was available.

Eligible patients entered the study and continued with the dose regimens of PEG-IFN alfa-2a and ribavirin they were taking prior to enrolment into the trial up to Week 24 of treatment. Patients who achieved at least a 2-log10 drop of HCV RNA at Week 12 (as compared to HCV RNA levels prior to treatment initiation) or had HCV RNA <15 IU/mL, and who were still taking study medication at treatment Week 24, were randomized at treatment Week 24 to one of the two study groups. Upon randomization, participants either stopped treatment (equaling 24 weeks of treatment) or continued treatment for another 24 weeks (equaling 48 weeks of treatment). A treatment free follow-up period of 24 weeks (for participants in the 48-week treatment group) or 48 weeks (participants in the 24-week treatment group) completed the study.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* serological evidence of chronic hepatitis C (CHC);
* CHC genotype 2 or 3;
* receiving PEGASYS + Copegus according to local standard of care and no rapid viral response (RVR);
* compensated liver disease.

Exclusion Criteria:

* pegylated interferon, standard interferon or ribavirin therapy at any time prior to initiation of current therapy with PEGASYS + Copegus;
* coinfection with hepatitis A or B, or human immunodeficiency virus (HIV);
* history or other evidence of decompensated liver disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2008-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (89):
- United States (35):
  - Birmingham, Alabama
  - La Jolla, California
  - Lancaster, California
  - Long Beach, California
  - Los Angeles, California
  - Sacramento, California
  - San Diego, California
  - Torrance, California
  - Aurora, Colorado
  - Jacksonville, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Honolulu, Hawaii
  - Baton Rouge, Louisiana
  - Opelousas, Louisiana
  - Boston, Massachusetts
  - Tupelo, Mississippi
  - St Louis, Missouri
  - Egg Harbour Township, New Jersey
  - Hackensack, New Jersey
  - Albuquerque, New Mexico
  - New York, New York
  - Syracuse, New York
  - Asheville, North Carolina
  - Chapel Hill, North Carolina
  - Winston-Salem, North Carolina
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Kingsport, Tennessee
  - Fort Sam Houston, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Fairfax, Virginia
  - Richmond, Virginia
- Australia (5):
  - Darlinghurst
  - Fremantle
  - Melbourne
  - Nedlands
  - Sydney
- Austria (5):
  - Graz
  - Innsbruck
  - Linz
  - Oberndorf
  - Vienna
- Belgium (5):
  - Antwerp
  - Brussels
  - Ghent
  - Kortrijk
  - Liège
- Brazil (10):
  - Brasília
  - Campinas
  - Porto Alegre
  - Ribeirão Preto
  - Rio de Janeiro
  - Santo André
  - São Luís
  - São Paulo
  - Sorocaba
  - Vitória
- Canada (4):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Hamilton, Ontario
  - Mississauga, Ontario
- Germany (16):
  - Berlin
  - Bonn
  - Cologne
  - Düsseldorf
  - Frankfurt am Main
  - Freiburg im Breisgau
  - Giessen
  - Hamburg
  - Heidelberg
  - Jena
  - Kiel
  - Mainz
  - München
  - Offenburg
  - Tübingen
  - Ulm
- Mexico (4):
  - Guadalajara
  - Mexicali
  - Mexico City
  - Puebla City
- Santurce, Puerto Rico
- Switzerland (4):
  - Lausanne
  - Lugano
  - Sankt Gallen
  - Zurich

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with Chronic Hepatitis C, Genotype 2 or 3 who had started therapy with PEG-IFN alfa-2a plus ribavirin according to local standard of care during a pre-study run-in phase and did not achieve a rapid viral response defined as HCV RNA <15 IU/mL at Week 4 of treatment were eligible and entered the screening phase between treatment Weeks 4-8.
Pre-assignment Details: 235 patients enrolled and continued with the dose regimens they were taking prior to enrolment up to Week 24 of treatment. Patients who achieved at least a 2-log10 drop of HCV RNA at Week 12 (compared to HCV RNA prior to treatment initiation) or had HCV RNA <15 IU/mL and who were still taking study medication at Week 24, were randomized at Week 24.
Groups:
- PEG-IFN Alfa-2a + Ribavirin for 24 Weeks: After 24 weeks of treatment with pegylated-interferon (peginterferon) alfa-2a (PEG-IFN alfa-2a) 180 μg/week plus ribavirin 800-1200 mg/day participants who achieved at least a 2-log10 drop of hepatitis C virus (HCV) ribonucleic acid (RNA) at Week 12 (as compared to HCV RNA levels prior to treatment initiation) or had HCV RNA <15 IU/mL, and who were still taking study medication at treatment Week 24 were randomized into the study, at which time treatment was stopped. Participants were followed for an additional 48 weeks during the treatment-free follow-up period.
Period: Treatment Period
Arm/Group | PEG-IFN Alfa-2a + Ribavirin for 24 Weeks | PEG-IFN Alfa-2a + Ribavirin for 48 Weeks
Started | 95 | 93
Completed | 95 (Patients who completed 24 weeks of treatment) | 66 (Patients who completed 48 weeks of treatment)
Not Completed | 0 | 27
Not completed — Adverse event/intercurrent illness | 0 | 9
Not completed — Death | 0 | 1
Not completed — Did not cooperate / refused treatment | 0 | 13
Not completed — Insufficient therapeutic response | 0 | 2
Not completed — Other | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Follow-up Period
Arm/Group | PEG-IFN Alfa-2a + Ribavirin for 24 Weeks | PEG-IFN Alfa-2a + Ribavirin for 48 Weeks
Started | 95 | 93
Completed | 66 (Patients who had an HCV RNA sample at 48 weeks of follow-up) | 78 (Patients who had an HCV RNA sample at 24 weeks of follow-up)
Not Completed | 29 | 15
Not completed — Relapse post-treatment | 11 | 3
Not completed — Failure to return | 10 | 2
Not completed — Patient withdrew consent | 5 | 4
Not completed — HCV-RNA detectable at end of treatment | 2 | 1
Not completed — Did not cooperate | 0 | 3
Not completed — Reason not specified | 1 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- PEG-IFN Alfa-2a + Ribavirin for 24 Weeks: After 24 weeks of treatment with peginterferon alfa-2a (PEG-IFN alfa-2a) 180 μg/week plus ribavirin 800-1200 mg/day participants who achieved at least a 2-log10 drop of hepatitis C virus (HCV) ribonucleic acid (RNA) at Week 12 (as compared to HCV RNA levels prior to treatment initiation) or had HCV RNA <15 IU/mL, and who were still taking study medication at treatment Week 24 were randomized into the study, at which time treatment was stopped. Participants were followed for an additional 48 weeks during the treatment-free follow-up period.
- Total: Total of all reporting groups
Arm/Group | PEG-IFN Alfa-2a + Ribavirin for 24 Weeks | PEG-IFN Alfa-2a + Ribavirin for 48 Weeks | Total
Number analyzed (Participants) | 95 | 93 | 188
Age Continuous [Mean (Standard Deviation); unit: years] | 48.8 (9.83) | 48.6 (10.12) | 48.7 (9.95)
Age, Customized [Number; unit: participants]
  ≤ 50 years | 47 | 53 | 100
  > 50 years | 48 | 40 | 88
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 39 | 79
  Male | 55 | 54 | 109
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian or white | 82 | 81 | 163
  Black | 8 | 6 | 14
  Asian or oriental | 1 | 2 | 3
  Other | 4 | 4 | 8
Hepatitis C virus (HCV) genotype [Number; unit: participants]
  HCV Genotype 2 | 19 | 19 | 38
  HCV Genotype 3 | 76 | 74 | 150
Pre-treatment HCV ribonucleic acid (RNA) [Mean (Standard Deviation); unit: log10 IU/mL] | 6.11 (0.624) | 6.17 (0.773) | 6.14 (0.700)
Region [Number; unit: participants] — Region (US and non-US) was used for stratification.
  participants
    Non-U.S. | 85 | 82 | 167
    U.S. | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Sustained Virologic Response 24 Weeks After Scheduled Completion of Treatment
Description: Sustained virological response (SVR) is defined as a single last HCV RNA measurement <15 IU/ml (measured using the Roche COBAS AmpliPrep / COBAS TaqMan HCV Test) 24 weeks after scheduled treatment completion, defined as Week 44 or later for participants randomized to the 24-week treatment period or Week 68 or later for participants randomized to the 48-week treatment period.
  Participants without measurements at the end of the 24-week untreated follow-up period were considered non-responders in the analysis.
Time Frame: 24 weeks after scheduled treatment completion (approximately Week 48 for participants in the 24-week treatment group and Week 72 for participants in the 48-week treatment group.
Population: All randomized patients.
Measure: Number; unit: percentage of participants
Arm/Group | PEG-IFN Alfa-2a + Ribavirin for 24 Weeks | PEG-IFN Alfa-2a + Ribavirin for 48 Weeks
Number analyzed (Participants) | 95 | 93
percentage of participants | 52 | 57
Statistical Analysis 1: Comparison: PEG-IFN Alfa-2a + Ribavirin for 24 Weeks vs PEG-IFN Alfa-2a + Ribavirin for 48 Weeks; In order to detect an improvement in SVR rate across all strata equivalent to an odds ratio of 2 (i.e. an increase in SVR by 15 to 16 percentage points at a power of 80% and a two-sided significance level of 0.05, 160 patients per treatment group (320 patients in total) were required; Test type: Superiority or Other; p = 0.4557, Cochran-Mantel-Haenszel; Stratified by HCV genotype (2 vs 3), region (US vs non-US) and initial Ribavirin dose (800mg vs 1000-1200mg); Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.45 to 1.43] — The odds ratio is the ratio of the odds of a response in the 24-week treatment group to the odds of a response in the 48-week treatment group. (second column)

2. Secondary Outcome: Percentage of Participants With Virological Response 72 Weeks After Treatment Initiation
Description: Virological response 72 weeks after treatment initiation is defined as the percentage of participants with HCV RNA <15 IU/mL as measured by the Roche COBAS AmpliPrep / COBAS TaqMan® HCV Test at 48 weeks post completion of the 24 week treatment period and 24 weeks post completion of the 48 week treatment period.
  Participants without Week 72 measurements were considered non-responders in the analysis.
Time Frame: Week 72
Population: All randomized patients.
Measure: Number; unit: percentage of participants
Arm/Group | PEG-IFN Alfa-2a + Ribavirin for 24 Weeks | PEG-IFN Alfa-2a + Ribavirin for 48 Weeks
Number analyzed (Participants) | 95 | 93
percentage of participants | 44 | 57
Statistical Analysis 1: Comparison: PEG-IFN Alfa-2a + Ribavirin for 24 Weeks vs PEG-IFN Alfa-2a + Ribavirin for 48 Weeks; Test type: Superiority or Other; p = 0.0788, Cochran-Mantel-Haenszel; Stratified by HCV genotype (2 vs 3), region (US vs non-US) and initial Ribavirin dose (800mg vs 1000-1200mg); Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.33 to 1.06] — The odds ratio is the ratio of the odds of a response in the 24-week treatment group to the odds of a response in the 48-week treatment group

3. Secondary Outcome: Percentage of Participants With Virological Response at End of Treatment
Description: Virological response at the end of treatment was defined as the percentage of participants with HCV RNA <15 IU/mL as measured by the Roche COBAS AmpliPrep / COBAS TaqMan® HCV Test after the last dose of study medication.
Time Frame: End of Treatment (Week 24 and Week 48 for each treatment group respectively).
Population: All randomized patients. A backward imputation approach was used when the HCV RNA measurement at end of treatment was missing and HCV RNA was <15 IU/mL at the first measurement after the end of treatment time window (the patient was regarded as having virological response at end of treatment).
Measure: Number; unit: percentage of participants
Arm/Group | PEG-IFN Alfa-2a + Ribavirin for 24 Weeks | PEG-IFN Alfa-2a + Ribavirin for 48 Weeks
Number analyzed (Participants) | 95 | 93
percentage of participants | 93 | 90
Statistical Analysis 1: Comparison: PEG-IFN Alfa-2a + Ribavirin for 24 Weeks vs PEG-IFN Alfa-2a + Ribavirin for 48 Weeks; Test type: Superiority or Other; p = 0.5654, Cochran-Mantel-Haenszel; Stratified by HCV genotype (2 vs 3), region (US vs non-US) and initial Ribavirin dose (800mg vs 1000-1200mg); Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.48 to 3.87] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Percentage of Participants With Virological Relapse
Description: Virological relapse defined as the percentage of participants with a virological response at end of treatment but who did not have a sustained virological response 24 weeks after the end of treatment.
  Virological response at end of treatment is defined as a single last HCV RNA measurement <15 IU/ml measured using the Roche COBAS AmpliPrep / COBAS TaqMan HCV Test at the day of last dose of study medication.
  Sustained virological response 24 weeks after the actual treatment end (SVR24) is defined as a single last HCV RNA measurement <15 IU/ml at least 20 weeks after treatment end.
Time Frame: End of treatment (Weeks 24 or 48) and 24 weeks after the end of treatment (weeks 48 and 72 in each treatment group respectively).
Population: Randomized patients with virological response at the end of treatment and at least one post-treatment HCV RNA measurement.
Measure: Number; unit: percentage of participants
Arm/Group | PEG-IFN Alfa-2a + Ribavirin for 24 Weeks | PEG-IFN Alfa-2a + Ribavirin for 48 Weeks
Number analyzed (Participants) | 83 | 80
percentage of participants | 41 | 29

5. Primary Outcome: Percentage of Participants With a Sustained Virologic Response 24 Weeks After Actual End of Treatment
Description: Sustained virological response (SVR) is defined as a single last HCV RNA measurement <15 IU/ml (measured using the Roche COBAS AmpliPrep / COBAS TaqMan HCV Test) at 24 weeks after actual end of study treatment. For participants in the 48-week treatment group who stopped study treatment prior to Week 48 for any reason, the HCV RNA measurements 24 weeks after actual end of treatment were used in the analysis. Participants without a 24-week post treatment measurement are considered non-responders.
Time Frame: 24 weeks after actual end of treatment (range from Week 48 to Week 72).
Population: All randomized patients.
Measure: Number; unit: percentage of participants
Arm/Group | PEG-IFN Alfa-2a + Ribavirin for 24 Weeks | PEG-IFN Alfa-2a + Ribavirin for 48 Weeks
Number analyzed (Participants) | 95 | 93
percentage of participants | 52 | 61
Statistical Analysis 1: Comparison: PEG-IFN Alfa-2a + Ribavirin for 24 Weeks vs PEG-IFN Alfa-2a + Ribavirin for 48 Weeks; Test type: Superiority or Other; p = 0.1934, Cochran-Mantel-Haenszel; Stratified by HCV genotype (2 vs 3), region (US vs non-US) and initial Ribavirin dose (800mg vs 1000-1200mg); Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.38 to 1.21] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Percentage of Participants With a Sustained Virologic Response 12 Weeks After Actual End of Treatment
Description: Sustained virological response (SVR) is defined as a single last HCV RNA measurement <15 IU/ml (measured using the Roche COBAS AmpliPrep / COBAS TaqMan HCV Test) at 12 weeks after actual end of study treatment. For participants in the 48-week treatment group who stopped study treatment prior to Week 48 for any reason, the HCV RNA measurements 12 weeks after actual end of treatment were used in the analysis. Participants without a 12-week post treatment measurement are considered non-responders.
Time Frame: 12 weeks after actual end of treatment (range from Week 36 to Week 60)
Population: All randomized patients.
Measure: Number; unit: percentage of participants
Arm/Group | PEG-IFN Alfa-2a + Ribavirin for 24 Weeks | PEG-IFN Alfa-2a + Ribavirin for 48 Weeks
Number analyzed (Participants) | 95 | 93
percentage of participants | 52 | 61
Statistical Analysis 1: Comparison: PEG-IFN Alfa-2a + Ribavirin for 24 Weeks vs PEG-IFN Alfa-2a + Ribavirin for 48 Weeks; Test type: Superiority or Other; p = 0.1934, Cochran-Mantel-Haenszel; Stratified by HCV genotype (2 vs 3), region (US vs non-US) and initial Ribavirin dose (800mg vs 1000-1200mg); Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.38 to 1.21] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as a sign or symptom, including intercurrent illness, that occurred during the course of the clinical study after treatment had started. A related AE is an event assessed by the Investigator to be remotely, possibly, or probably related to study treatment according to criteria provided in the protocol. A severe AE was an event graded by the Investigator as "incapacitating with inability to work or perform normal daily activity". A serious AE (SAE) was defined as any experience that suggests a significant hazard, contraindication, side effect or precaution. This includes any experience which was fatal; was life-threatening; required inpatient hospitalization or prolongation of an existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/ birth defect; was medically significant or required intervention to prevent one or other of the outcomes listed above.
Time Frame: From Week 1 through Week 72.
Measure: Number; unit: participants
Arm/Group | PEG-IFN Alfa-2a + Ribavirin for 24 Weeks | PEG-IFN Alfa-2a + Ribavirin for 48 Weeks
Number analyzed (Participants) | 95 | 93
participants
  Any AE | 81 | 88
  Severe AE | 13 | 24
  AE related to PEG-IFN alfa-2a | 78 | 86
  AE related to ribavirin | 72 | 83
  Serious AE | 4 | 11
  SAE related to PEG-IFN alfa-2a | 0 | 7
  SAE related to ribavirin | 0 | 4
  Deaths | 0 | 1

ADVERSE EVENTS:
Time Frame: 72 weeks.
Arm/Group | PEG-IFN Alfa-2a + Ribavirin for 24 Weeks | PEG-IFN Alfa-2a + Ribavirin for 48 Weeks
Serious Adverse Events (participants affected / at risk) | 4/95 | 11/93
Other Adverse Events (participants affected / at risk) | 81/95 | 87/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-IFN Alfa-2a + Ribavirin for 24 Weeks (N=95) | PEG-IFN Alfa-2a + Ribavirin for 48 Weeks (N=93)
Psychotic disorder (Psychiatric disorders) | 0 | 1
Alcohol abuse (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Mesangioproliferative glomerulonephritis (Renal and urinary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-IFN Alfa-2a + Ribavirin for 24 Weeks (N=95) | PEG-IFN Alfa-2a + Ribavirin for 48 Weeks (N=93)
Fatigue (General disorders) | 33 | 47
Asthenia (General disorders) | 18 | 14
Pyrexia (General disorders) | 11 | 11
Influenza like illness (General disorders) | 14 | 7
Irritability (General disorders) | 12 | 4
Chills (General disorders) | 1 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 17 | 20
Alopecia (Skin and subcutaneous tissue disorders) | 15 | 17
Dry skin (Skin and subcutaneous tissue disorders) | 13 | 14
Rash (Skin and subcutaneous tissue disorders) | 8 | 9
Nausea (Gastrointestinal disorders) | 13 | 24
Diarrhoea (Gastrointestinal disorders) | 7 | 14
Abdominal pain upper (Gastrointestinal disorders) | 7 | 8
Dyspepsia (Gastrointestinal disorders) | 2 | 10
Abdominal pain (Gastrointestinal disorders) | 3 | 5
Vomiting (Gastrointestinal disorders) | 3 | 5
Dry mouth (Gastrointestinal disorders) | 2 | 5
Insomnia (Psychiatric disorders) | 21 | 21
Depression (Psychiatric disorders) | 13 | 11
Sleep disorder (Psychiatric disorders) | 6 | 6
Anxiety (Psychiatric disorders) | 5 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 3
Headache (Nervous system disorders) | 17 | 30
Dizziness (Nervous system disorders) | 6 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Anaemia (Blood and lymphatic system disorders) | 8 | 9
Neutropenia (Blood and lymphatic system disorders) | 7 | 7
Decreased appetite (Metabolism and nutrition disorders) | 8 | 15
Weight decreased (Investigations) | 7 | 9
Hypertension (Vascular disorders) | 2 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.